CLINICAL TRIAL: NCT02235805
Title: The Effects of Magnesium on Vascular Stiffness: A Long-term Study in Healthy Overweight and Slightly Obese Men and Women
Brief Title: Magnesium and Vascular Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MEC 14-3-021
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Metabolic Syndrome; Obesity; Magnesium Supplementation; Vascular Stiffness; Vascular Function
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium Citrate (Experimental)
  Interventions: Dietary Supplement: Magnesium Citrate
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate — One capsule thrice daily that contains magnesium citrate (total daily dose: 350 mg elemental magnesium) at breakfast, lunch and dinner for 24 weeks
  Arms: Magnesium Citrate
Dietary Supplement: Placebo — One capsule thrice daily that contains placebo at breakfast, lunch and dinner for 24 weeks
  Arms: Placebo

SUMMARY:
Observational epidemiologic studies have observed an inverse relationship between daily dietary magnesium intake and blood pressure (BP). Except for BP, magnesium may also beneficially affect other cardiovascular risk markers. Whether all these effects translate into improved vascular function is not known. Different vascular function markers at various stages on the pathway between diet and disease exist. One of these markers, vascular stiffness, is closely related to the process of atherosclerosis, an independent cardiovascular risk factor, and predictive of future cardiovascular events and mortality. To examine the integrated effects of interventions on cardiovascular risk, vascular stiffness may therefore serve as a marker at the later stage of cardiovascular disease development.

Therefore, it is imperative to examine in a 24-week, randomized, double-blind, placebo-controlled, two-way parallel-group human intervention study, the effect of magnesium on vascular stiffness. Focus will be on carotid-femoral pulse wave velocity (PWV), the gold standard for the evaluation of vascular elasticity, to quantify vascular stiffness. Urinary excretion of magnesium will be used to assess dietary magnesium uptake. Furthermore, time courses of an increased magnesium intake on changes in BP, other markers reflecting vascular function, and plasma biomarkers related to low-grade inflammation and vascular activity will be measured to unravel possible cause-effect relationships.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 45-70 years
* Women postmenopausal: two or more years after last menstruation
* BMI between 25-35 kg/m2 (overweight and slightly obese)
* Plasma glucose < 7.0 mmol/L
* Serum total cholesterol < 8.0 mmol/L
* Serum triacylglycerol < 4.5 mmol/L
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Less than 21 alcoholic consumptions per week
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of proton pump inhibitors or medication known to treat blood pressure, serum lipid or glucose metabolism
* No use of dietary supplements or an investigational product within another biomedical within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebro vascular accident
* Willingness to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* High habitual dietary magnesium intake
* Plasma glucose ≥ 7.0 mmol/L
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.5 mmol/L
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 21 alcoholic consumptions per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use of proton pump inhibitors or medication known to treat blood pressure, serum lipid or glucose metabolism
* Use of dietary supplements or an investigational product within another biomedical within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebro vascular accident
* Not willing to give up being a blood donor (or having donated blood) from 8 weeks before the start of the study and during the study
* Not or difficult to venipuncture as evidenced during the screening visit

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Vascular stiffness: effects of magnesium citrate supplementation | Baseline (0 weeks) and after medium-term (12 weeks) and long-term (24 weeks) magnesium citrate supplementation
  Carotid-femoral pulse wave velocity (PWV)

SECONDARY OUTCOMES:
Vascular function markers: effects of magnesium citrate supplementation | Baseline (0 weeks) and after long-term (24 weeks) magnesium citrate supplementation
  Flow-mediated dilation (FMD) of the brachial artery, pulse wave analysis (PWA) (also at 12 weeks), peripheral arterial tonometry (PAT) and retinal microvascular diameters (also at 12 weeks)
Metabolic risk markers related to the metabolic syndrome: effects of magnesium citrate supplementation | Baseline (0 weeks) and after medium-term (12 weeks) and long-term (24 weeks) magnesium citrate supplementation
  Biomarkers for low-grade inflammation and endothelial activation
Blood pressure: effects of magnesium citrate supplementation | Baseline (0 weeks) and after long-term (24 weeks) magnesium citrate supplementation
  Office (also at 12 weeks) and 24-hour ambulatory blood pressure

OTHER OUTCOMES:
Dietary magnesium uptake | Baseline (0 weeks) and after long-term (24 weeks) magnesium citrate supplementation
  24-hour urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Schutten JC, Joris PJ, Minovic I, Post A, van Beek AP, de Borst MH, Mensink RP, Bakker SJL. Long-term magnesium supplementation improves glucocorticoid metabolism: A post-hoc analysis of an intervention trial. Clin Endocrinol (Oxf). 2021 Feb;94(2):150-157. doi: 10.1111/cen.14350. Epub 2020 Oct 26. PMID 33030273
- [Derived] Joris PJ, Plat J, Bakker SJ, Mensink RP. Long-term magnesium supplementation improves arterial stiffness in overweight and obese adults: results of a randomized, double-blind, placebo-controlled intervention trial. Am J Clin Nutr. 2016 May;103(5):1260-6. doi: 10.3945/ajcn.116.131466. Epub 2016 Apr 6. PMID 27053384